CLINICAL TRIAL: NCT01016379
Title: Genome-Wide Interrogations in Childhood Acute Lymphoblastic Leukemia (ALL)
Brief Title: Studying DNA in Blood and Bone Marrow Samples From Young Patients With Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL08B2; COG-AALL08B2; CDR0000659101; NCI-2011-02200 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood and Bone Marrow
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Other: biologic sample preservation procedure
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how well patients will respond to treatment.

PURPOSE: This research study is looking at DNA in blood and bone marrow samples from young patients with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To manage and oversee determination of genome-wide genotypes using common laboratory methodologies for young patients with newly diagnosed acute lymphoblastic leukemia (ALL).
* To provide a mechanism for storing, distributing, and tracking usage of blast and germline genomic information for approved projects.
* To facilitate research for childhood ALL using genome-wide germline and blast data to identify genetic variations associated with important phenotypes: treatment response (e.g., relapse risk, minimal residual disease status), adverse effects (e.g., osteonecrosis, infection risk, neurotoxicity), risk of ALL, and risk of ALL subtypes (e.g., TEL/AML1, BCR/ABL, T-cell).
* To provide a data resource, that can be linked with additional tumor cell information, to better characterize the biology and subtypes of childhood ALL.

OUTLINE: This is a multicenter study.

DNA from previously collected and banked blood and bone marrow samples is utilized for genome-wide genotyping.

Genotype data is only used to examine specific questions related to the epidemiology and etiology of leukemia, response of leukemia to treatment, risk of recurrence, risk for development of side effects, and complications related to treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute lymphoblastic leukemia (ALL)
* Previously enrolled in COG-9900, COG-C1991, COG-AALL03B1, COG-AALL05B1, COG-AALL08P1, or other current COG or legacy trials for ALL AND consented to submit blood and marrow samples for biological research studies
* Meets ≥ 1 of the following criteria:

  * Germline DNA that has been extracted from blood (preferentially) or bone marrow (if no appropriate blood available) that was collected on or after Day 28 of remission indication therapy, or is known to come from a sample that contained < 10% leukemic blasts
  * ALL blast DNA that has been extracted from bone marrow (preferentially) or blood (if from a sample that contained > 90% leukemic blasts and no diagnostic bone marrow is available) that was collected at the time of ALL diagnosis

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Young Patients With Acute Lymphoblastic Leukemia
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Determination of genome-wide genotypes
Mechanism for storing, distributing, and tracking usage of blast and germline genomic information
Identification of genetic variations associated with important phenotypes (treatment response, adverse effects, risk of acute lymphoblastic leukemia [ALL], and risk of ALL subtypes)
Data resource, that can be linked with additional tumor cell information, to better characterize the biology and subtypes of childhood ALL

CONTACTS AND LOCATIONS:
Overall Officials: Mignon Loh, MD, Study Chair — University of California, San Francisco